CLINICAL TRIAL: NCT00061165
Title: Obesity Prevention in African American School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPAASC (completed)
Record Dates: First submitted 2003-05-21; First posted 2003-05-23 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: obesity; overweight; children; adolescents; African American; diet; nutrition; physical activity; Chicago
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Schools; Exercise

INTERVENTIONS:
Behavioral: School + family changes promoting healthy eating + activity

SUMMARY:
Obesity is the second leading preventable cause of disease and death in the United States. Low socioeconomic status (SES) and minorities are disproportionately affected. Obesity prevention among children and adolescents is a public health priority. Schools have been identified as key settings for obesity prevention; however, most health education interventions have had only a moderate effect on body weight. We propose a randomized intervention trial (pilot study) to test the feasibility and effectiveness of a school-based, environmental obesity prevention program in urban low-SES African American students. Schools, students and their families, and local communities will be involved to promote healthy eating and physical activity (HEPA) for prevention of childhood obesity. Six Chicago public schools will be randomly assigned as intervention (4 schools) and controls (2 schools). Focus group studies will assess needs and barriers for promotion of HEPA and guide the intervention. The intervention group will receive a School Environment Enrichment (SEE) program to modify the school physical and social environment, targeting food service, recess, physical education (PE) and school climate, and a Community Support & Environment Modification (CSEM) program, involving local corner and chain grocery stores to promote healthy eating among students and their families. Family involvement will be included for 5th and 6th graders, who will be followed for two years, to test ways to modify family environment. To assess the intervention effectiveness, multilevel data will be collected from schools (eg, food service, recess and PE), students (eg, body weight, eating and physical activity), parents (eg, family food purchasing practices) and communities (eg, available choices of snack foods in local stores). In addition, process evaluation data will be collected to assess the feasibility and acceptance (participation and satisfaction) of various intervention components by the target audience. The primary outcome variable is change in students' body weight status; secondary outcomes include changes in students' eating behavior and physical activity and changes in target environmental factors. In addition, cost-effectiveness of the intervention will be determined. If the intervention proves effective, a full-scale study will be developed. Findings from this study will provide insights into the prevention of obesity among low-SES and minority students.

ELIGIBILITY:
All 4-6th graders in the selected public schools in Chicago and their parents/guardians

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Youfa Wang, PhD, MD — University of Illinois at Chicago, Department of Human Nutrition
Locations (1):
- University of Illinois at Chicago, Department of Human Nutrition, Chicago, Illinois, United States